

Status: Approved, Version: 5.0 Approved Date: 26 Aug 2021



## Device Protocol for CLU484-P002 / NCT05010512 Title: Clinical Performance of Two Commercial, Daily Disposable Contact Lenses

Protocol Number: CLU484-P002

Clinical Investigation

Type:

Postmarket Interventional / Confirmatory

DAILIES TOTAL1® contact lenses (delefilcon A) Test Product:

Alcon Research, LLC, and its affiliates ("Alcon") Sponsor Name and Address:

6201 South Freeway

Fort Worth, Texas 76134-2099

Property of Alcon Confidential May not be used, divulged, published, or otherwise disclosed without the consent of Alcon

Document ID: V-CLN-0010987


Status: Approved, Version: 5.0 Approved Date: 26 Aug 2021

#### Investigator Agreement:

- I have read the clinical study described herein, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practices; applicable international and national regulations, laws, guidelines, and standards; the conditions of approval imposed by the reviewing IRB or regulatory authority; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current investigator's brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authority? | | | |
|---|---|---|---|---|
| | □ No | □Yes | | |
| | Have you ever been involved in a study or other research that was terminated? | | | |
| | □ No | □Yes | | |
| | If yes, ple | ease explair | n here: | |
| Pr | incipal inv | estigator: | | |
| | | | Signature | Date |
| | ame and prosition: | ofessional | | |
| A | ddress: | | | |
| Ph | one Numb | er: | | |
| | Off-hours Emergency<br>Phone Number: | | | |

## **Table of Contents**

| De | vice Prote | ocol for CLU484-P002 | 1 |
|---|---|---|---|
| Ta | ble of Co | ntents | 3 |
| Lis | st of Table | es | 5 |
| Lis | st of Figu | res | 6 |
| 1 | GLOSS | ARY OF TERMS | 7 |
| 2 | LIST OF | F ACRONYMS AND ABBREVIATIONS | 14 |
| 3 | PROTO | COL SUMMARY | 15 |
| 4 | PROTO | COL AMENDMENTS | 22 |
| 5 | INTROI | DUCTION | 23 |
| | 5.1 | Rationale and Background | |
| | 5.2 | Purpose of the Study | |
| | 5.3 | Risks and Benefits | |
| 6 | STUDY | OBJECTIVES | 24 |
| | 6.1 | Primary Objective(s) | 24 |
| | 6.2 | Secondary Objective(s) | 25 |
| | 6.4 | Safety Objective(s) | |
| 7 | INVES 7 | TIGATIONAL PLAN | 26 |
| | 7.1 | Study Design. | 26 |
| | 7.2 | Rationale for Study Design. | 27 |
| | | 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design Adaptations | 27 |
| | 7.3 | Rationale for Duration of Treatment/Follow-Up | |
| | 7.4 | Rationale for Choice of Comparator Product | |
| | 7.5 | Data Monitoring Committee | 28 |
| 8 | STUDY | POPULATION | 28 |
| | 8.1 | Inclusion Criteria | 28 |
| | 8.2 | Exclusion Criteria | 29 |
| | 8.3 | Rescreening of Subjects | 30 |
| 9 | TREATI | MENTS ADMINISTERED | 30 |

| | 9.1 | Investigational Product(s) | 30 |
|---|---|---|---|
| | 9.2 | Other Medical Device or Medication Specified for Use During the Study | 34 |
| | 9.3 | Treatment Assignment / Randomization | 34 |
| | 9.4 | Treatment masking | 35 |
| | 9.5 | Accountability Procedures | 37 |
| | 9.6 | Changes to concomitant medications, treatments/ procedures | 37 |
| 10 | STUDY | PROCEDURES AND ASSESSMENTS | |
| | 10.1 | Informed Consent and Screening | 38 |
| | 10.2 | Description of Study Procedures and Assessments | |
| | | 10.2.1 Demographics | |
| | | 10.2.2 Medical History | |
| | | 10.2.3 Investigational Product compliance | 39 |
| | | 10.2.4 Adverse Event Collection: Safety Assessment | 39 |
| | | 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment | 39 |
| | | 10.2.6 Device Deficiencies: Safety Assessment | 39 |
| | 10.3 | Unscheduled Visits | 39 |
| | 10.4 | Discontinued Subjects | 40 |
| | | 10.4.1 Screen Failures | 40 |
| | | 10.4.2 Discontinuations | 40 |
| | | 10.4.3 Schedule of Procedures and Assessments for Subjects | |
| | | Discontinued from Investigational Product | |
| | 10.5 | Clinical Study Termination | 41 |
| | | 10.5.1 Follow-up of subjects after study participation has ended | 41 |
| 11 | ADVER | SE EVENTS AND DEVICE DEFICIENCIES | 42 |
| | 11.1 | General Information | 42 |
| | 11.2 | Monitoring for Adverse Events | 44 |
| | 11.3 | Procedures for Recording and Reporting | 45 |
| | 11.4 | Return product analysis (if applicable) | 47 |
| | 11.5 | Unmasking of the Study Treatment | 47 |
| | 11.6 | Follow-Up of Subjects with Adverse Events | 47 |
| | 11.7 | Pregnancy in the Clinical Study | 48 |
| 12 | ANALY | SIS PLAN | 48 |
| | 12.1 | Subject Evaluability | 48 |

Table 2–1

Status: Approved, Version: 5.0 Approved Date: 26 Aug 2021

| | 12.2 | Analysis Sets | 48 |
|----|--------|------------------------------------------------------|----|
| | | 12.2.1 Safety Analysis Set | 48 |
| | | 12.2.2 Full Analysis Set | 49 |
| | 12.3 | Demographic and Baseline Characteristics | |
| | 12.4 | Effectiveness Analyses | |
| | | 12.4.1 Analysis of Primary Effectiveness Endpoint(s) | |
| | | 12.4.1.1 Statistical Hypotheses | |
| | | 12.4.1.2 Analysis Methods | 50 |
| | 12.5 | Handling of Missing Data | 53 |
| | 12.6 | Safety Analyses | 53 |
| | 12.7 | Interim Analyses and Reporting | 54 |
| | 12.8 | Sample Size Justification | 54 |
| 13 | DATA H | ANDLING AND ADMINISTRATIVE REQUIREMENTS | 55 |
| | 13.1 | Subject Confidentiality | 55 |
| | 13.2 | Completion of Source Documents and Case Report Forms | 55 |
| | 13.3 | Data Review and Clarifications | 56 |
| | 13.4 | Sponsor and Monitoring Responsibilities | 56 |
| | 13.5 | Regulatory Documentation and Records Retention | 57 |
| | 13.6 | Quality Assurance and Quality Control | 57 |
| 14 | ETHICS | | 58 |
| 15 | REFERE | ENCES | 59 |
| | 15.1 | Regulations and Standards | 59 |
| | 15.2 | Scientific and Other References | |
| | | List of Tables | |

| Document ID:<br>V-CLN-001098 | Status: Approved, Version: 5.0 Approved Date: 26 Aug 2021 | |
|---|---|---|
| Table 3–1 | Schedule of Study Procedures and Assessments | 20 |
| Table 6–1 | Primary Objective(s) | 24 |
| Table 6–3 | Safety Objective(s) | 25 |
| Table 9–1 | Test Product | 30 |
| Table 9–2 | Comparator Product | 32 |
| | List of Figures | |
| Figure 11-1 | Categorization of All Adverse Events | 42 |

## 1 GLOSSARY OF TERMS

| Names of test product(s) | Throughout this document, test product(s) will be referred to as: DAILIES TOTAL1® contact lenses (DT1). |
|---|---|
| Name of Comparator | Throughout this document, comparator product(s) will be |
| Product(s) | referred to as: BAUSCH+LOMB INFUSE <sup>™</sup> contact lenses (Infuse) |
| Adverse Device Effect | Adverse event related to the use of an investigational |
| (ADE) | medical device or comparator. |
| | Note: This definition includes adverse events resulting from |
| | insufficient or inadequate instructions for use, deployment, |
| | implantation, installation, or operation; any malfunction; |
| | and use error or intentional misuse. |
| Adverse Event (AE) | Untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device or comparator and whether anticipated or unanticipated. Note: For subjects, this definition includes events related to |
| | the investigational medical device, comparator, or the |
| | procedures involved. For users or other persons, this |
| | definition is restricted to the use of investigational medical |
| | device or comparator. |
| | Requirements for reporting Adverse Events in the study can |
| | be found in Section 11. |
| Anticipated Serious | An effect which by its nature, incidence, severity, or |
| Adverse Device Effect | outcome has been identified in the risk assessment. |
| (ASADE) | |

| Clinical Investigation Plan (CIP) | The document(s) stating the rationale, objectives, design, and prespecified analysis, methodology, organization, monitoring, conduct, and record-keeping of the clinical investigation. Note: The protocol and other documents referenced in the protocol (for example, the Statistical Analysis Plan, the Manual of Procedures, the Deviations and Evaluability Plan, and the Protocol Monitoring Plan) comprise the CIP. |
|---|---|
| Clinical Investigation | The document describing the design, execution, statistical |
| Report (CIR) / Clinical | analysis, and results of a clinical investigation. The Clinical |
| Study Report | Investigation Report is synonymous with the Clinical Study Report. |
| Device Deficiency | Inadequacy of a medical device with respect to its identity, quality, durability, reliability, usability, safety, or performance. |
| | Note: This definition includes malfunctions, use errors, and inadequacy in the information supplied by the manufacturer including labelling related to the investigational medical device or the comparator. |
| | Requirements for reporting Device Deficiencies in the study can be found in Section 11. |
| Enrolled Subject | Any subject who signs an informed consent form for participation in the study. |
| Point of Enrollment | The time at which, following recruitment and before any clinical investigation-related procedures are undertaken, a |
| | subject signs and dates the informed consent form. |

| T 1 | |
|---|---|
| Interventional Clinical Trial | A pre- or postmarket clinical investigation where the assignment of a subject to a particular medical device is |
| | decided in advance by a clinical investigation plan, or |
| | diagnostic or monitoring procedures requested in the CIP are |
| | in addition to those available as normal clinical practice and |
| | burden the subject. |
| Investigational Product | A preventative (vaccine), a therapeutic (drug or biologic), |
| | device, diagnostic, or palliative used as a test or comparator |
| | product in a clinical trial, including a product with a |
| | marketing authorization when used or assembled |
| | (formulated or packaged) in a way different from the |
| | authorized form, or when used for an unauthorized |
| | indication, or when used to gain further information about |
| | the authorized form. |
| 25.40 | |
| Malfunction | Failure of an investigational medical device to perform in |
| | accordance with its intended purpose when used in |
| | accordance with the instructions for use or clinical |
| | investigation plan (CIP), or investigator's brochure (IB). |
| Noninterventional Study | Clinical investigation that draws inferences about the |
| | possible effect of an intervention on subjects, but the |
| | investigator has not assigned subjects into intervention |
| | groups based on a protocol and has not made any attempts to |
| | collect data on variables beyond those available throughout |
| | the course of normal clinical practice and burden to the |
| | subject. |
| | NOTE: The term "noninterventional" is synonymous with |
| | "observational." |
| Nonserious Adverse Event | Adverse event that does not meet the criteria for a serious adverse event. |

| Postmarketing / | Any study conducted within the conditions laid down in |
|---|---|
| Postauthorization study | product labelling and other conditions laid down for the |
| | marketing of the product or under normal conditions of use. |
| | A postmarketing study falls either within the definitions of |
| | an interventional or a noninterventional study and may also |
| | fall within the definition of a postapproval study. |
| Product Complaint | Any oral, electronic, or written communication that alleges |
| | deficiencies related to the identity (labeling), quality, |
| | durability, reliability, safety, effectiveness, or performance |
| | of a marketed product, including failure of the product, |
| | labeling, or packaging to meet specifications, whether or not |
| | the product is related to or caused the alleged deficiency. A |
| | complaint may allege that an adverse event or medical |
| | device malfunction has occurred. |
| Randomized Subject | Any subject who is assigned a randomized treatment. |
| Serious Adverse Device | Adverse device effect that has resulted in any of the |
| Effect (SADE) | consequences characteristic of a serious adverse event. |

## Serious Adverse Event (SAE)

Adverse event that led to any of the following:

- Death.
- A serious deterioration in the health of the subject, users or other persons as defined by one or more of the following:
  - a) a life-threatening illness or injury

    Note: Life-threatening means that the individual was

    at immediate risk of death from the event as it

    occurred, i.e., it does not include an event which

    hypothetically might have caused death had it

    occurred in a more severe form.
  - b) any potentially sight-threatening event or permanent impairment to a body structure or a body function including chronic diseases.
  - c) inpatient hospitalization or prolonged hospitalization.
  - d) a medical or surgical intervention to prevent a) or b).
  - e) any indirect harm as a consequence of incorrect diagnostic test results when used within manufacturer's instructions for use.
- Fetal distress, fetal death, congenital abnormality or birth defect including physical or mental impairment.

Note: Planned hospitalization for a preexisting condition, or a procedure required by the CIP, without serious deterioration in health, is not considered a serious adverse event.

Refer to Section 11 for additional SAEs.

| Serious Health Threat | Signal from any adverse event or device deficiency that indicates an imminent risk of death or a serious deterioration in the health in subjects, users, or other persons, and that requires prompt remedial action for other subjects, users, or other persons. Note: This would include events that are of significant and unexpected nature such that they become alarming as a potential serious health hazard or possibility of multiple deaths occurring at short intervals. |
|---|---|
| Study Start | The start of the study is considered to coincide with the enrollment of the first patient. |
| Study Completion | The completion of the study is considered to coincide with the study-level last subject last visit or the decision to terminate the trial, whichever is later. |
| Unanticipated Serious Adverse Device Effect (USADE) | Serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the risk assessment. |
| Use Error | User action or lack of user action while using the medical device that leads to a different result than that intended by the manufacturer or expected by the user. Note: a) Use error includes the inability of the user to complete a task. b) Use errors can result from a mismatch between the characteristics of the user, user interface, task, or use environment. c) Users might be aware or unaware that a use error has occurred. d) An unexpected physiological response of the patient is not by itself considered a use error. e) A malfunction of a medical device that causes an unexpected result is not considered a use error." |

| Vulnerable Subject | An individual who is unable to fully understand all aspects |
|---|---|
| | of the investigation that are relevant to the decision to |
| | participate, or who could be manipulated or unduly |
| | influenced as a result of a compromised position, |
| | expectation of benefits or fear of retaliatory response. |

## 2 LIST OF ACRONYMS AND ABBREVIATIONS

Table 2–1 List of Acronyms and Abbreviations Used in This Protocol

| Abbreviation | Definition |
|--------------|------------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| CFR | Code of Federal Regulations |
| CIP | Clinical Investigation Plan |
| CIR | Clinical Investigation Report |
| CRF | Case report form |
| CTT | Clinical Trial Team |
| D | Diopter |
| DEP | Deviations and evaluability plan |
| DFU | Directions for use |
| DT1 | DAILIES TOTAL1® contact lenses |
| eCRF | Electronic case report form |
| EDC | Electronic Data Capture |
| GCP | Good Clinical Practice |
| IB | Investigator's brochure |
| ICF | Informed consent form |
| Infuse | BAUSCH+LOMB INFUSE <sup>™</sup> contact lenses |
| IP | Investigational product |
| IRB | Institutional review board |
| ISO | International Organization for Standardization |
| LID | Lens Identification Number |
| LogMAR | Logarithm of the minimum angle of resolution |
| mm | Millimeter |
| MOP | Manual of procedures |
| N/A | Not applicable |
| NI | Noninferiority |
| PI | Principal investigator |
| SD | Standard deviation |
| SADE | Serious adverse device effect |
| SAE | Serious adverse event |
| SLE | Slit lamp examination |
| SOP | Standard operating procedure |
| T2B | Top-2-Box |
| US | United States |
| VA | Visual acuity |
| VAS | Visual Analog Scale |

## **3 PROTOCOL SUMMARY**

| Investigational Device | |
|---|---|
| product type | |
| product type | |
| Study type Interventional | |
| Investigational Test Product: DT1 contact lenses | |
| Products Comparator Product: Infuse contact lenses | |
| Purpose and To compare the clinical performance of DT1 contact lenses | s with |
| Scientific Rationale Infuse contact lenses | |
| for the Study | |
| Objective(s) The primary objective of this study is to demonstrate | |
| noninferiority (NI) in visual acuity (VA) at distance when | wearing |
| DT1 contact lenses compared to Infuse contact lenses. | 8 |
| Endpoint(s) Primary Effectiveness | |
| Distance VA (logMAR) with study lenses | |



| | Safety |
|---|---|
| | Biomicroscopy |
| | Adverse Events |
| | Device deficiencies |
| Study Design | This will be a prospective, randomized, |
| | , controlled, double-masked, crossover, daily |
| | wear clinical study. Subject participation in the study will be |
| | approximately 3 weeks with 16-22 days of lens wear. |
| | DT1 (T) 0 ( 0 ( 12 ) 1 |
| | DT1 (Test): 8 (-0/+3) days |
| | Infuse (Comparator): 8 (-0/+3) days |
| Subject population | Planned number of subjects enrolled/consented: ~110 |
| | Planned number of completed subjects: 100 |
| G'4 1T 4' | DI 1 1 C 1: 1 1: 0 |
| Sites and Locations | Planned number of clinical sites: ~ 8 |
| | Planned locations (initial list of locations, which may change |
| | during start up or conduct according to study needs): United States |

| Key inclusion criteria (See Section 8.1 for a complete list of inclusion criteria) | <ul> <li>Habitual soft contact lens wearers in both eyes, aged 18 or over who have at least 3 months of contact lens wearing experience, and who wear their habitual lenses at least 5 days per week and at least 10 hours per day.</li> <li>To qualify, subjects must have a manifest refraction of ≤ 0.75 D in each eye, and a BCVA (with manifest refraction) better than or equal to 20/25 (Snellen) or 0.10 (logMAR) in each eye</li> </ul> | | |
|---|---|---|---|
| Key exclusion criteria (See Section 8.2 for a complete list of exclusion criteria) Data analysis and sample size justification | <ul> <li>Current/previous DT1 and Infuse habitual lens wearers and any monovision &amp; multifocal lens wearers.</li> <li>Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.</li> <li>Planned Data Analysis</li> <li>To address the primary and key exploratory effectiveness objectives, planned analyses are summarized below:</li> </ul> | | |
| | Endpoint Primary Distance VA | DT1 vs Infuse Noninferiority | Mixed effect repeated measures NI margin = 0.05 (logMAR) |



Table 3-1 Schedule of Study Procedures and Assessments

| Visit | Visit 1 Screening/Baseline/ Dispense Lens 1 | Visit 2<br>Week 1 Follow-<br>up Lens 1 /<br>Dispense Lens 2 | Visit 3<br>Week 1<br>Follow-up<br>Lens 2 / Exit | Early Exit | Unscheduled Visit |
|---|---|---|---|---|---|
| | | 8 (-0/+3) days after<br>Visit 1 | 8 (-0/+3) days<br>after Visit 2 | N/A | N/A |
| Informed Consent | X | | | | |
| Demographics | X | | | | |
| Medical History | X | X | X | X | X |
| Concomitant<br>Medications‡ | X | X | X | X | X |
| Inclusion/Exclusion | X | | | | |
| Habitual lens information (brand, power) | X | | | | |
| VA with habitual<br>correction (OD, OS,<br>LogMAR distance)* | X | | X (Exit<br>procedure) | X | (X) |
| Manifest refraction and<br>BCVA with manifest<br>refraction (OD, OS,<br>logMAR distance) * | X | (X) | (X) | (X) | (X) |
| Biomicroscopy | X | X | X | X | X |
| Trial lens fitting (DT1 and Infuse) | Х | | | | |
| Randomize | X | | | | |
| Dispense (provide) study lenses* | X | Х | | | (X) |

Document ID: V-CLN-0010987

| Visit | Visit 1 Screening/Baseline/ Dispense Lens 1 | Visit 2<br>Week 1 Follow-<br>up Lens 1 /<br>Dispense Lens 2 | Visit 3<br>Week 1<br>Follow-up<br>Lens 2 / Exit | Early Exit | Unscheduled Visit |
|---|---|---|---|---|---|
| | | 8 (-0/+3) days after<br>Visit 1 | 8 (-0/+3) days<br>after Visit 2 | N/A | N/A |
| VA (logMAR distance)<br>with study lenses, OD,<br>OS | | X | X | (X) | (X) |

| Visit | Visit 1 Screening/Baseline/ Dispense Lens 1 | Visit 2<br>Week 1 Follow-<br>up Lens 1 /<br>Dispense Lens 2 | Visit 3<br>Week 1<br>Follow-up<br>Lens 2 / Exit | Early Exit | Unscheduled Visit |
|---|---|---|---|---|---|
| | | 8 (-0/+3) days after<br>Visit 1 | 8 (-0/+3) days<br>after Visit 2 | N/A | N/A |
| AEs | X | X | X | X | X |
| Device Deficiencies | X | X | X | X | X |
| Exit Form | (X) | (X) | X | X | (X) |

(X) assessment performed as necessary, e.g., decrease of VA by 2 lines or more with investigational product (IP)



#### 4 PROTOCOL AMENDMENTS

Modification of the protocol is prohibited without prior written agreement in the form of a protocol amendment. All amendments must be created by the study sponsor and must be approved by the IRB/IEC and global and regional Health Authorities, as applicable, prior to implementation except when required to mitigate immediate safety risks or when the changes involve only logistical or administrative revisions.

Amendments may necessitate that the informed consent and other study-related material be revised. If the consent form is revised, all subjects currently enrolled in the study must sign the approved, revised informed consent (re-consent), as required by the IRB/IEC.

#### 5 INTRODUCTION

#### 5.1 Rationale and Background

It is estimated that soft contact lenses account for over 90% of lens fits. Moreover, almost 32% of soft contact lenses were prescribed in a daily disposable modality. DT1 contact lenses were introduced as a unique dual technology that combines a low water content silicone hydrogel core, to achieve optimal oxygen supply, with a high water content hydrogel surface to provide a highly lubricious, wettable lens. Previous studies support the hypothesis that Water Gradient Technology in DT1 lenses produces superior clinical performance and subjective acceptance.

## 5.2 Purpose of the Study

The purpose of this study is to evaluate the overall clinical performance of DT1contact lenses when compared to another commercially available daily disposable contact lens, Infuse.

| The design of this study is justified based upon preclinical and clinical testing, as described within the package insert. Infuse contact lenses were chosen as the comparator product because these lenses have the same wear modality. |
|---|
| At the end of the study, a clinical study report will be prepared in accordance with applicable regulatory requirements and standards. |

#### 5.3 Risks and Benefits

The clinical investigation process risks are managed through appropriate training and monitoring according to the protocol-specific monitoring plan. Investigational device risks, including risks associated with use of device and methods and procedures for application of device, are defined in the product labeling and are managed through review of safety assessments outlined in this protocol.

Contact lenses may offer improved peripheral vision and the convenience of not wearing spectacles. Material properties and design characteristics of the contact lens in development are features consistent with successful contact lens wear.

The test products are for daily wear use under a daily disposable wear modality; further details on any known potential risks and benefits can be found in the package insert. The test products are not intended for use with a cleaning/disinfecting solution, and the biocompatibility with lens care solutions and any associated clinical effects are unknown.

A summary of the known potential risks and benefits associated with the DT1 and Infuse contact lenses can be found in the package insert. Risks are minimized by compliance with the eligibility criteria and study procedures, and through close supervision by a licensed clinician during exposure to the study lenses

#### 6 STUDY OBJECTIVES

## 6.1 Primary Objective(s)

Table 6–1 Primary Objective(s)

| Objective(s) | Endpoint(s) |
|---|---|
| Demonstrate noninferiority in the VA at | |
| distance when wearing DT1 contact lenses | Distance VA (locMAD) with study longer |
| compared to Infuse contact lenses. | Distance VA (logMAR) with study lenses |

## 6.2 Secondary Objective(s)

Not Applicable



## 6.4 Safety Objective(s)

Table 6–3 Safety Objective(s)

Objective(s) Endpoint(s)

Duty of care and evaluation of safety profile AEs of the investigational products. Biomicroscopy findings Device deficiencies

#### 7 INVESTIGATIONAL PLAN

#### 7.1 Study Design

This will be a prospective, randomized, \_\_\_\_\_\_\_, controlled, double-masked, crossover, daily wear clinical study. Subject participation in the study will be approximately 3 weeks with approximately 16-22 days of lens wear.



## 7.2 Rationale for Study Design

This study design is justified based upon an evaluation of the results of relevant preclinical and clinical testing, as described within the package inserts.

| The crossover design will ensure that the same subject is exposed to both the test and |
|---|
| comparator lens materials; |
| study will include only those |
| subjects who are current wearers of spherical soft contact lenses in both eyes with at least 3 |
| months wearing experience, with a minimum wearing time of 5 days per week and 10 hours |
| per day. |
| Furthermore, the subjects will not be permitted to use lubrication/rewetting drops during the |
| duration of the study as this may confound the primary effectiveness endpoint. The study will |
| exclude any habitual DT1 and Infuse contact lens wearers in the past 3 months prior to |
| consent in order to reduce potential bias of wearers to their habitual contact lenses. The study |
| will also exclude subjects who wish to wear their contact lenses in monovision modality |
| during the study and multifocal lens wearers. |
| 7.2.1 Purpose and Timing of Interim Analyses and Resulting Design |
| Adaptations |
| An interim analysis will not be performed. |
| 7.3 Rationale for Duration of Treatment/Follow-Up |
| Subjects will wear each study product bilaterally for approximately 1 week. |
| The primary |
| will be assessed on approximately after 1 week of wearing each study product |

## 7.4 Rationale for Choice of Comparator Product

B+L Infuse spherical, daily disposable contact lenses were chosen as the comparator product because these lenses have the same wear modality and replacement schedule

## 7.5 Data Monitoring Committee

Not Applicable

#### 8 STUDY POPULATION

The study population consists of male and female subjects (18 years or older) with a diagnosis of refractive ametropia (myopia and hyperopia)It is aimed to enroll (consent) approximately 110 subjects in approximately 8 sites throughout the United States, with a target of 100 total subjects completed, with 13 (intended minimum) to 14 (maximum) subjects per site. Site-specific targets may vary based upon individual site capabilities. Estimated time needed to recruit subjects for the study is approximately 4 weeks; however, unanticipated circumstances may shorten or lengthen this time and would not require amendment of this protocol. Because a 10% screening failure rate is expected, approximately 110 subjects are expected to be enrolled.

#### 8.1 Inclusion Criteria

Written informed consent must be obtained before any study specific assessment is performed. Upon signing informed consent, the subject is considered enrolled in the study.

Subjects eligible for inclusion in this study must fulfill all of the following criteria:

- 1 Subject must be at least 18 years of age.
- 2 Subject must be able to understand and must sign an ICF that has been approved by an IRB.
- 3 Successful wear of spherical soft contact lenses in both eyes for a minimum of 5 days per week and 10 hours per day during the past 3 months.
- 4 Manifest cylinder  $\leq 0.75$  D in each eye.
- 5 BCVA (with manifest refraction) better than or equal to 0.10 (logMAR) in each eye.





#### 8.2 Exclusion Criteria

Subjects fulfilling any of the following criteria are not eligible for participation in this study.

1 Current/previous DT1and Infuse habitual lens wearers and any monovision & multifocal lens wearers.



Wearing habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.



## 8.3 Rescreening of Subjects

Rescreening of subjects is not allowed in this study.

#### 9 TREATMENTS ADMINISTERED

## 9.1 Investigational Product(s)

Test Product(s): DAILIES TOTAL1 contact lenses

Comparator Product(s) (If

Infuse contact lenses

applicable):

Table 9–1 Test Product

| Test Product | DAILIES TOTAL1 contact lenses (DT1) |
|---|---|
| Manufacturer | Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, Texas 76134-2099 USA |
| Indication for use and intended purpose in the current study | The intended use of this contact lens is for vision correction. |

| Product description | Material: delefilcon A |
|---|---|
| and parameters | Water content: 33% |
| available for this | |
| study | • Power range: -1.00 to -6.00 D, 0.25 D steps |
| Study | Base curve (mm): 8.5 The state of the |
| | • Diameter (mm): 14.1 |
| Formulation | Refer to package insert |
| Usage | • Wear: |
| | o Daily Wear |
| | o Bilateral |
| | Replacement period: Daily Disposable |
| | Exposure: Approximately 10 hours per day, every day over an |
| | 8-11 day period |
| | • Lens Care: N/A |
| Number/Amount of | At the dispense visit, sites will ensure that subjects are given |
| product to be | adequate lenses to last until the next planned study visit, allowing |
| provided to the | for planned and unplanned lens replacements. |
| subject | for planned and anplanned tens replacements. |
| Packaging | Blister foil pack |
| description | |
| Labeling description | Lens Foil label includes: |
| | • lens identifier |
| | base curve |
| | diameter |
| | <ul> <li>packing solution</li> </ul> |
| | • power |
| | • lot number |
| | expiration date |
| | • content statement |
| | <ul> <li>investigational device statement</li> </ul> |
| | <ul> <li>sponsor information</li> </ul> |
| | • sponsor information |

| | country of origin |
|---|---|
| | • Provided in packages of approximately 12 lenses per power, |
| | identified with the following: |
| | - a color coded label stating the protocol number |
| | - lens identifier |
| | - power |
| | - an investigational use only statement |
| | - tracking number |
| Storage conditions | Lenses should be stored at room temperature |
| Additional | N/A |
| information | |
| Supply | Fitting sets will be provided by the sponsor before the start of |
| | the study to be used during Visit 1. Fitting sets will include |
| | sphere powers ranging from -1.00 to -6.00D, in -0.25D steps. |
| | • Small inventories of each power will be provided for dispense to subjects at Visit 1. If needed, additional IP can be ordered and provided upon request. |
| | Refer to the MOP for a detailed description |

Table 9–2Comparator Product

| Comparator | Infuse contact lenses (Infuse) |
|---|---|
| Product(s) | |
| Manufacturer | Bausch + Lomb |
| Indication for Use | The intended use of this contact lens is for vision correction |
| Product description | Material: kalifilcon A |
| and parameters<br>available for this<br>study | • Water content: 45% |
| | • Power range: -1.00 to -6.00 D, in 0.25 D steps |
| | • Base curve (mm): 8.6 |
| | • Diameter (mm): 14.2 |
| Formulation | Refer to package insert |
| Usage | • Wear: |

| | <ul> <li>Daily Wear</li> <li>Bilateral</li> <li>Replacement period: Daily Disposable</li> <li>Exposure: Approximately 10 hours per day, every day over an 8-11 day period</li> <li>Lens Care: N/A</li> </ul> |
|---|---|
| Number/Amount of Product to be Provided to the subject | At the dispense visit, sites will ensure that subjects are given adequate lenses to last until the next planned study visit, allowing for planned and unplanned lens replacements. |
| Packaging description | Blister foil pack |
| Labeling description | Lenses have investigational labeling, which includes: lens identifier |

| | - tracking number |
|---|---|
| Storage conditions | Lenses should be stored at room temperature |
| Additional identifying information | N/A |
| Supply | <ul> <li>Fitting sets will be supplied in packages of 12 per power, ranging from -1.00 to -6.00D, in -0.25D steps.</li> <li>Small inventories of each power will be provided for dispense to subjects at Visit 1. If needed, additional IP can be provided upon request.</li> <li>Refer to the MOP for a detailed description</li> </ul> |

More information on the test product can be found in the Package Inserts.

# 9.2 Other Medical Device or Medication Specified for Use During the Study

No other medical devices or medications are required to be used in conjunction with the treatments during the clinical study.

## 9.3 Treatment Assignment / Randomization

Subjects will be randomized in a 1:1 manner to receive one of 2 lens sequences:

| Sequence | EDC/randomization integration system | Lens Name |
|------------|--------------------------------------|------------|
| Sequence 1 | | DT1/Infuse |
| Sequence 2 | | Infuse/DT1 |

Only after signing the ICF, a subject will be assigned a subject number by the electronic data capture system.

A randomization list will be generated using a validated system that automates the random assignment of treatment (lens sequence) to randomization numbers in the specified ratio.

Subjects will be assigned treatment (lens sequence) according to the randomization list uploaded in the randomization system. The randomization list will be generated and maintained by the study sponsor.

At Visit 1, all eligible subjects will be randomized via the EDC/randomization integration system to one of the treatments (lens sequences). The investigator's delegate will access the respective system after confirming that the subject meets all the eligibility criteria. A randomization number will be automatically assigned to the subject according to the subject randomization list but will not be communicated to the site user. The EDC/randomization integration system will inform the site user of the treatment (lens sequence) assignment to be dispensed to the subject.

#### 9.4 Treatment masking

This study is double-masked. All members associated with the study (at the site and the study sponsor) are masked to the assigned treatment





This level of masking will be maintained throughout the conduct of the study. Unmasking will occur only after all planned study data have been validated, and the database locked.

Masked study personnel must avoid seeking information that may compromise masking.

In the event of a medical emergency where the knowledge of subject treatment is required, an individual investigator will have the ability to unmask the treatment assignment for a specific subject after contacting an appropriate study sponsor representative if time allows.
## 9.5 Accountability Procedures

Upon receipt of the IPs, the investigator or delegate must conduct an inventory.

Throughout the study, the investigator or delegate must maintain records of IP dispensation and collection for each subject. This record must be made available to the study monitor for the purposes of verifying the accounting of IP supplies. Any discrepancies and/or deficiencies between the observed disposition and the written account must be recorded along with an explanation. All IPs sent to the investigator must be accounted for by study sponsor personnel, and in no case be used in an unauthorized situation.

The investigator should make every effort to collect unused lenses, foils, and supplies from subjects.

It is the investigator's responsibility to ensure that:

- All study products are accounted for and not used in any unauthorized manner
- All unused products are available for return to the study sponsor, as directed
- Any study lenses associated with a device deficiency or with any product-related adverse
  event (i.e., ADE or SADE) are returned to the study sponsor for investigation, unless
  otherwise directed by the sponsor. Refer to Section 11 of this protocol for additional
  information on the reporting of device deficiencies and AEs and the return of study
  products associated with these events.

The investigator is responsible for proper disposition of all unused IPs at the conclusion of the study, according to the instructions provided in the MOP.

# 9.6 Changes to concomitant medications, treatments/ procedures

After the subject is enrolled into the study, the investigator must instruct the subject to notify the study site about:

- Any new medications
- Alterations in dose or dose schedules for current medications,
- Any medical procedure or hospitalization that occurred or is planned
- Any nondrug therapies (including physical therapy and blood transfusions).

The investigator must document this information in the subject's case history source documents.

#### 10 STUDY PROCEDURES AND ASSESSMENTS

#### 10.1 Informed Consent and Screening

The investigator or delegate must explain the purpose and nature of the study, and have the subject read, sign, and date the IRB/IEC-approved informed consent document. The subject must sign the ICF BEFORE any study-specific procedures or assessments can be performed, including study-specific screening procedures. Additionally, have the individual obtaining consent from the subject and a witness, if applicable, sign and date the informed consent document.

The investigator or delegate must provide a copy of the signed document to the subject and place the original signed document in the subject's chart, or provide documentation as required by local regulations.

#### 10.2 Description of Study Procedures and Assessments

Detailed descriptions of assessments and procedures are provided in the MOP. The investigator is responsible for ensuring responsibilities for all procedures and assessments are delegated to appropriately qualified site personnel.

# 10.2.1 Demographics

Obtain demographic information including age, race, ethnicity, and sex.

# **10.2.2** Medical History

Collect medical history information, including information on all medications used within the past 30 days. Include herbal therapies, vitamins, and all over-the-counter as well as prescription medications. Throughout the subject's participation, obtain information on any changes in medical health and/or the use of concomitant medications.

Medical History and Concomitant Medications will be collected in the eCRF as outlined in the MOP.

## 10.2.3 Investigational Product compliance

Review subject compliance with the IP usage and adjunct product usage and collect all used and unused study IPs and other products that were dispensed.

## 10.2.4 Adverse Event Collection: Safety Assessment

Assess and record any adverse events that are observed or reported since the previous visit, including those associated with changes in concomitant medication dosing.

## 10.2.5 Slit Lamp Biomicroscopy: Safety Assessment

SLE of the cornea, iris/anterior chamber and lens must be performed in both eyes before instillation of any diagnostic eye drops.

## 10.2.6 Device Deficiencies: Safety Assessment

Assess and record any Device Deficiencies that are reported or observed since the previous visit. Requirements for reporting device deficiencies in the study can be found in Section 11.

#### 10.3 Unscheduled Visits

If a subject visit occurs between any regularly scheduled visit and the visit is conducted by study personnel, this visit must be documented as an Unscheduled Visit. If the subject seeks medical attention outside the clinic (for example, at an Emergency Room) or at the clinic but is seen by nonstudy personnel, the investigator is to capture adverse event-related information on the Adverse Event form upon becoming aware.

During all unscheduled visits, the investigator must conduct the following procedures:

- Collect Adverse Event information
- Record changes in medical condition or concomitant medication

The investigator may perform additional procedures for proper diagnosis and treatment of the subject. The investigator must document this information in the subject's case history source documents.

If during an Unscheduled Visit the subject is discontinuing the IP or discontinuing from the study, the investigator must conduct Exit procedures according to Table 3–1 Schedule of Study Procedures and Assessments, as possible.

## 10.4 Discontinued Subjects

#### **10.4.1 Screen Failures**

Subjects who were excluded from the study after signing the informed consent and prior to randomization to product/dispense of study product.

The investigator must document the reason for screen failure in the subject's case history source documents.

Subject numbers must not be re-used.

#### 10.4.2 Discontinuations

Discontinued subjects are individuals who voluntarily withdraw or are withdrawn from the study by the investigator after signing the informed consent.

Subject numbers of discontinued subjects must not be re-used (i.e., subject replacement is not allowed).

Subjects may discontinue from study or study treatment at any time for any reason. Subjects may also be discontinued from study treatment at any time if, in the opinion of the investigator, continued treatment poses a risk to their health.

For subjects discontinuing from the study, the investigator must complete all Exit procedures according to Table 3–1 Schedule of Study Procedures and Assessments, if the subject is willing and able, and if in the opinion of the investigator it is safe for the subject to do so.

The investigator must document the reason for study or treatment discontinuation in the subject's case history source documents.

To ensure the safety of all subjects who discontinue early, investigators must assess each subject and, if necessary, advise them of any therapies and/or medical procedures that may be needed to maintain their health.

# 10.4.3 Schedule of Procedures and Assessments for Subjects Discontinued from Investigational Product

Other than screen failures, if a subject discontinues from the study, the subject should undergo an Early Exit Visit. Refer to Table 3–1

## 10.5 Clinical Study Termination

The study sponsor reserves the right to suspend or close the investigational site or suspend or terminate the study in its entirety at any time.

If the clinical study is prematurely terminated or suspended by the study sponsor:

- The study sponsor must:
  - Immediately notify the investigator(s) and subsequently provide instructions for study termination.
  - o Inform the investigator and the regulatory authorities of the termination/suspension and the reason(s) for the termination/suspension.
- The investigator must:
  - Promptly notify the IRB/IEC of the termination or suspension and of the reasons.
  - Provide subjects with recommendations for poststudy treatment options as needed.

The investigator may terminate the site's participation in the study for reasonable cause.

# 10.5.1 Follow-up of subjects after study participation has ended

Following this study, the subject will return to their eye care professional for their routine eye care.



#### 11 ADVERSE EVENTS AND DEVICE DEFICIENCIES

#### 11.1 General Information

An AE is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users, or other persons, whether or not related to the investigational medical device (test product). Refer to the Glossary of Terms and figures below for categories of AEs and SAEs.

Figure 11-1 Categorization of All Adverse Events



Figure 11-2 Categorization of All Serious Adverse Events



#### **Specific Events Relevant to this Protocol**

#### Serious Adverse Events

In addition to reporting all AEs (serious and nonserious) meeting the definitions, the investigator must report any occurrence of the following as an SAE:

- An ocular infection including a presumed infectious ulcer with any of the following characteristics:
  - Central or paracentral location
  - Penetration of Bowman's membrane
  - o Infiltrates > 2 mm diameter
  - Iritis
  - Increase in intraocular pressure
  - Culture positive for microorganisms
  - Increasing size or severity at subsequent visits
- Any central or paracentral corneal event (such as neovascularization) that results in permanent opacification
- Hypopyon

Document ID: V-CLN-0010987

Status: Approved, Version: 5.0 Approved Date: 26 Aug 2021

- Hyphema
- Neovascularization within the central 6 mm of the cornea
- Permanent vision loss as defined by loss of 2 or more lines of BCVA from enrollment visit that fails to resolve
- Uveitis (anterior, intermediate, or posterior)
- Corneal abrasion affecting  $\geq 50\%$  of corneal surface area

#### **Device Deficiencies**

A device deficiency is inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance. A device deficiency may or may not be associated with patient harm (i.e., ADE or SADE); however, not all ADEs or SADEs are due to a device deficiency. The investigator should determine the applicable category listed in the Device Deficiency eCRF for the identified or suspect device deficiency and report any patient harm separately. Examples of device deficiencies include the following:

- Failure to meet product specifications (e.g., incorrect lens power/diameter/base curve/color)
- Lens/solution cloudy
- Lens surface/edge defect
- Torn lens during handling/in pack
- Packaging deficit (e.g., mislabeled product, tampered seal, leaking bottle/container)
- Suspect product contamination
- Lack of performance

## 11.2 Monitoring for Adverse Events

At each visit, after the subject has had the opportunity to spontaneously mention any problems, the investigator should inquire about AEs by asking the standard questions shown below and report as applicable:

- "Have you had any health problems since your last study visit?"
- "Have there been any changes in the medicines you take because of a new health issue since your last study visit?"

In addition, changes in *any protocol-specific parameters* evaluated during the study are to be reviewed by the investigator. Any untoward (unfavorable and unintended) change in *a protocol-specific parameter* that is clinically relevant, in the opinion of the investigator, is to be reported as an AE. These clinically relevant changes will be reported regardless of causality.

## 11.3 Procedures for Recording and Reporting

AEs are collected from the time of informed consent Any preexisting medical conditions or signs/symptoms present in a subject prior to the start of the study (i.e., before informed consent is signed) are not considered AEs in the study and should be recorded in the Medical History section of the eCRF.

In addition, temporary lens awareness or visual changes during the fitting process are not considered AEs if the investigator assesses that the symptom(s) can reasonably resolve within the anticipated adaptation period.

For each recorded event, the ADEs and SAEs documentation must include: date of occurrence, severity, treatment (if applicable), outcome, and assessments of the seriousness and causality. In addition, the investigator must document all device deficiencies reported or observed with test and comparator products on the Device Deficiency eCRF. The site must submit all available information on ADEs, SAEs, and device deficiencies to the study sponsor immediately as follows:

- All SAEs must be reported immediately (within 24 hours) of the investigator's or site's awareness.
- ADEs that do not meet seriousness criteria and device deficiencies must be reported within 10 calendar days of the Investigator's or site's awareness.
- A printed copy of the completed *Serious Adverse Event and Adverse Device Effect* and/or *Device Deficiency* eCRF must be included with product returns.
- Additional relevant information after initial reporting must be entered into the eCRF as soon as the data become available.
- Document any changes to concomitant medications on the appropriate eCRFs.
- Document all relevant information from Discharge Summary, Autopsy Report, Certificate of Death, etc., if applicable, in narrative section of the *Serious Adverse Event eCRF and Adverse Device Effect(for related AEs)* eCRF.

*Note:* Should the EDC system become nonoperational, the site must complete the appropriate paper Serious Adverse Event and Adverse Device Effect and/or Device Deficiency Form. The completed form is emailed to the study sponsor at msus.safety@alcon.com for US according to the timelines outlined above; however, the reported information must be entered into the EDC system once it becomes operational.

Study sponsor representatives may be contacted for any protocol-related question and their contact information is provided in the Manual of Procedures that accompanies this protocol.

Further, depending upon the nature of the AE or device deficiency being reported, the study sponsor may request copies of applicable portions of the subject's medical records. The investigator must also report all AEs and device deficiencies that could have led to a SADE according to the requirements of regulatory authorities or IRB/IEC.

#### **Intensity and Causality Assessments**

Where appropriate, the investigator must assess the intensity (severity) of the AE based on medical judgment with consideration of any subjective symptom(s), as defined below:

#### Intensity (Severity)

Mild An AE is mild if the subject is aware of but can easily tolerate the sign or

symptom.

Moderate An AE is moderate if the sign or symptom results in discomfort significant

enough to cause interference with the subject's usual activities.

Severe An AE is severe if the sign or symptom is incapacitating and results in the

subject's inability to work or engage in their usual activities.

For every AE in the study, the investigator must assess the causality (Related or Not Related to the medical device or study procedure). An assessment of causality will also be performed by study sponsor utilizing the same definitions, as shown below:

#### **Causality**

Related

An AE classified as related may be either definitely related or possibly related where a direct cause and effect relationship with the medical device or study procedure has not been demonstrated, but there is a reasonable possibility that the AE was caused by the medical device or study procedure.

Not Related An AE classified as not related may either be definitely unrelated or simply unlikely to be related (i.e., there are other more likely causes for the AE).

The study sponsor will assess the AEs and may upgrade the investigator's assessment of seriousness and/or causality. The study sponsor will notify the investigator of any AEs that is upgraded from nonserious to serious or from unrelated to related.

## 11.4 Return product analysis (if applicable)

Study sponsor representatives and their contact information are provided in the MOP that accompanies this protocol.

Alcon products associated with device deficiencies and/or product related AEs should be returned and must include the Complaint #, which will be provided by study sponsor after the case is entered in the study sponsor's Global Product Complaint Management System (GPCMS).

## 11.5 Unmasking of the Study Treatment

Masked information on the identity of the assigned medical device should not be disclosed during the study. If the treatment code needs to be broken in the interest of subject safety, the investigator is encouraged to contact an appropriate study sponsor representative prior to unmasking the information if there is sufficient time. Dependent upon the individual circumstances (i.e. medical emergency), the code may be broken prior to contact with the Study Sponsor. The Study Sponsor must be informed of all cases in which the code was broken and of the circumstances involved. Additionally, the Study Sponsor may be required to unmask the information in order to fulfill expedited regulatory reporting requirements

# 11.6 Follow-Up of Subjects with Adverse Events

The investigator is responsible for adequate and safe medical care of subjects during the study and for ensuring that appropriate medical care and relevant follow-up procedures are maintained after the study.

The investigator should provide the study sponsor with any new safety information (which includes new AEs and changes to previously reported AEs) that may affect the safety evaluation of the device. For AEs that are unresolved/ongoing at time of subject exit from study, any additional information received at follow-up should be documented in the eCRFs up to study completion (i.e., database lock).

All complaints received after this time period will be considered and processed as spontaneous (following the post- market vigilance procedures) and should be communicated to the medical device's manufacturer as per local requirements.

The investigator should also report complaints on non-Alcon products (i.e., Infuse contact lenses) directly to the manufacturer as per the manufacturer's instructions or local regulatory requirements.

## 11.7 Pregnancy in the Clinical Study

Women of childbearing potential or women who are pregnant at the time of study entry are not excluded from participation. Pregnancy should be included in the Medical History section of the eCRF when a pregnant woman enters the study or if a woman becomes pregnant during the study. Pregnancy is not reportable as an AE; however, complications may be reportable and will be decided on a case-by-case basis .An Alcon form will be utilized to capture all pregnancy- related information until birth of the child.

#### 12 ANALYSIS PLAN

Continuous variables will be summarized using the number of observations, mean, standard deviation (SD), median, minimum, and maximum, as well as confidence intervals (CIs) or confidence limits where applicable. Categorical variables will be summarized with frequencies and percentages from each category.

Any deviations to the analysis plan will be updated during the course of the study as part of a protocol amendment or will be detailed in the clinical study report.

# 12.1 Subject Evaluability

Final subject evaluability must be determined prior to breaking the code for masked treatment (lens sequence) assignment and locking the database, based upon the Deviations and Evaluability Plan (DEP).

# 12.2 Analysis Sets

# 12.2.1 Safety Analysis Set

Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. As such, the safety analysis set will include all subjects/eyes exposed to any study lenses

| 1 . 1. 1 1 | |
|---|---|
| evaluated in this study, | |
| For treat | ıtment- |
| emergent safety analyses, subjects/eyes will be categorized under the actual study len | ses |
| exposed in the corresponding lens sequence. | |
| 12.2.2 Full Analysis Set | |
| The full analysis set (FAS) is the set of all randomized subjects who are exposed to a | nv stud |

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study.

# 12.3 Demographic and Baseline Characteristics

Demographic information will be summarized by lens sequence and overall. Frequencies and percentages will be presented for categorical variables such as sex, age group, race, and ethnicity. Number of observations, mean, SD, median, minimum, and maximum will be presented for continuous variables such as age.

# 12.4 Effectiveness Analyses

| This study defines 1 primary, |
|---|
| will use the FAS as the primary analysis set. |
| The primary effectiveness endpoint of distance VA will be tested at one-sided $\alpha = 0.05$ for |
| noninferiority |

# 12.4.1 Analysis of Primary Effectiveness Endpoint(s)

The primary objective of this study is to demonstrate noninferiority in distance VA when wearing DT1 contact lenses compared to Infuse contact lenses. The primary endpoint is distance VA with study lenses, collected for each eye in logMAR.

## 12.4.1.1 Statistical Hypotheses

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.05 for noninferiority:

$$H_0$$
:  $\mu_{(T)} - \mu_{(C)} \ge 0.05$   
 $H_a$ :  $\mu_{(T)} - \mu_{(C)} < 0.05$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the mean distance VA for DT1 and Infuse, respectively, on the logMAR scale.

## 12.4.1.2 Analysis Methods

A mixed effect repeated measures model will be utilized to test these hypotheses. The model will include terms for lens, period, and sequence as fixed effects. Within-subject correlation due to eye and the crossover design will also be accounted for in the model. Lens difference (DT1 minus Infuse) and the corresponding one-sided 95% upper confidence limit will be computed. Noninferiority in distance VA will be declared if upper confidence limit is less than 0.05.



## 12.5 Handling of Missing Data

All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out

#### 12.6 Safety Analyses

The safety endpoints are:

- AEs
- Biomicroscopy findings
- Device Deficiencies

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of occurrence of adverse events as well as the other listed parameters.

All AEs occurring from the time a subject signs informed consent to study exit will be accounted for in the reporting. Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis. Descriptive summaries (frequencies and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities Preferred Terms. AEs leading to study discontinuation and SAEs will be identified. Individual subject listings will be provided, as necessary.

Individual subject listings will be provided for AEs that occur after signing informed consent but prior to exposure to IP.

Each biomicroscopy parameter will be tabulated by its grade. For each applicable biomicroscopy parameter, counts and percentages of eyes that experience an increase of  $\geq 2$  grades from baseline (last assessment prior to study lens exposure) to any subsequent visit within the same period will be presented. A supportive listing will be generated which will include all biomicroscopy data from all visits within the same period for those eyes experiencing the increase.

Two listings for device deficiencies, prior to exposure to study contact lenses and treatmentemergent, will be provided. Additionally, each device deficiency category will be tabulated.

No inferential testing will be conducted for the safety analyses.

## 12.7 Interim Analyses and Reporting

There are no plans to conduct an interim analysis and no criteria by which the study would be terminated early based upon statistical determination.

## 12.8 Sample Size Justification

Sample size calculation is based on a prior clinical study which evaluated performance of DT1 and Infuse.

#### **Primary Effectiveness**

To demonstrate noninferiority (margin = 0.05 in logMAR; ½ line in Snellen) in distance VA as a one-tailed hypothesis with  $\alpha$ =0.05, and using a standard deviation of 0.0497 for paired differences, 80% power can be attained with a sample size of 8 (4 per sequence).





#### 13 DATA HANDLING AND ADMINISTRATIVE REQUIREMENTS

## 13.1 Subject Confidentiality

The investigator must ensure that the subject's identity is kept confidential throughout the course of the study. In particular, the investigator must keep an enrollment log with confidential identifying information that corresponds to the subject numbers and initials of each study participant. The study sponsor may collect a copy of the enrollment log without any directly identifying subject information.

The study sponsor may share patient-level data collected in this trial with qualified researchers to help facilitate product development or enhancements in research that is not directly related to the study objectives. The Informed Consent explains this to the study subject.

# 13.2 Completion of Source Documents and Case Report Forms

The nature and location of all source documents will be identified to ensure that original data required to complete the CRFs exist and are accessible for verification by the site monitor, and all discrepancies shall be appropriately documented via the query resolution process. Site monitors are appointed by the study sponsor and are independent of study site staff.

If electronic records are maintained, the method of verification must be determined in advance of starting the study.

At a minimum, source documents include the following information for each subject:

- Subject identification (name, sex, race/ethnicity)
- Documentation of subject eligibility
- Date of informed consent
- Dates of visits
- Documentation that protocol specific procedures were performed
- Results of study parameters, as required by the protocol
- IP accountability records
- Documentation of AEs and other safety parameters (if applicable)
- Records regarding medical histories and the use of concomitant therapies prior to and during the study
- Date of study completion and reason for early discontinuation, if applicable

It is required that the author of an entry in the source documents be identifiable. Direct access to source documentation (medical records) must be allowed for the purpose of verifying that the data recorded on the CRF are consistent with the original source data.

Only designated individuals at the site will complete the CRFs. The CRFs must be completed at regular intervals following the clinical study visit schedule. It is expected that all data reported have corresponding entries in the source documents. The principal investigator is responsible for reviewing and certifying that the CRFs are accurate and complete. The only subject identifiers recorded on the CRFs will be subject number, and subject demographic information.

#### 13.3 Data Review and Clarifications

A review of CRF data to the subject's source data will be completed by the site monitor to ensure completeness and accuracy. After the CRFs have been completed, additional data clarifications and/or additions may be needed as a result of the data cleaning process. Data clarifications are documented and are part of each subject's CRF.

# 13.4 Sponsor and Monitoring Responsibilities

The study sponsor will select principal investigators that are qualified by education, training, and experience to assume responsibility for the proper conduct of this clinical trial.

The study sponsor is financially funding this clinical trial and will compensate the investigator and/or the Institution(s) at which the study is conducted in accordance with a signed clinical trial agreement.

The study sponsor will designate a monitor to conduct the appropriate site visits at the appropriate intervals according to the study monitoring plan. The clinical investigation will be monitored to ensure that the rights and well-being of the subjects are protected, the reported data are accurate, complete, and verifiable from the source documents, and the study is conducted in compliance with the current approved protocol (and amendments[s], if applicable), with current GCP, and with applicable regulatory requirements.

The site may not screen subjects or perform the informed consent process on any subject until it receives a notification from an appropriate study sponsor representative that the site may commence conducting study activities. Monitoring will be conducted periodically while the clinical study is ongoing. Monitoring methods may include site visits, telephone, written and fax correspondence. Close-out visits will take place after the last visit of the last subject at the site.

A coordinating investigator may be identified by the study sponsor to review and endorse the final study report. In cases where a coordinating investigator is engaged, the study sponsor will select the coordinating investigator based upon their experience, qualifications, active study participation, and their willingness and availability to take on this role.

# 13.5 Regulatory Documentation and Records Retention

The investigator is required to maintain up-to-date, complete regulatory documentation as indicated by the study sponsor and the investigator's files will be reviewed as part of the ongoing study monitoring. Financial information is to be kept separately.

Additionally, the investigator must keep study records and source documents consistent with the terms of the clinical study agreement with the study sponsor. If the investigator retires, relocates, or for any other reason withdraws from responsibility of keeping the study records, then the study sponsor must be notified and suitable arrangements made for retention of study records and source documents needed to comply with national and international regulations.

# 13.6 Quality Assurance and Quality Control

The study sponsor will secure agreement from all involved parties to ensure direct access to all study related sites, source data and documents, and reports for the purpose of monitoring and auditing by the study sponsor, and inspection by domestic and foreign regulatory

authorities. Quality control will be applied to each stage of data handling to ensure that all data are reliable and have been processed correctly. Agreements made by the study sponsor with the investigator/institution and any other parties involved in the clinical study will be provided in writing as part of the protocol or as a separate agreement.

#### 14 ETHICS

Investigations are conducted in compliance with Good Clinical Practices; international and national regulations, laws and guidelines; the conditions of approval imposed by reviewing IRBs/IECs or regulatory authorities; and in accordance with the ethical medical research principles outlined in the Declaration of Helsinki.

- The SOPs of the study sponsor and contract research organizations participating in the conduct of the clinical study and all other applicable regulations shall apply.
- Notifications and timelines for reporting protocol deviations should be based upon applicable Ethics Committee requirements.

The investigator must ensure that all personnel involved in the conduct of the study are qualified to perform their assigned responsibilities through relevant education, training, and experience. The investigator and all clinical study staff must conduct the clinical study in compliance with the protocol. Deviations from this protocol, regulatory requirements, and/or GCP must be recorded and reported to the Sponsor prior to database lock. If needed, corrective and preventive action should be identified, implemented, and documented within the study records. Use of waivers to deviate from the clinical protocol is prohibited.

Before clinical study initiation, this protocol, the informed consent form, any other written information given to subjects, and any advertisements planned for subject recruitment must be approved by an IRB/IEC. The investigator must provide documentation of the IRB/IEC approval to the study sponsor. The approval must be dated and must identify the applicable protocol, amendments (if any), informed consent form, assent form (if any), all applicable recruiting materials, written information for subject, and subject compensation programs. The IRB/IEC must be provided with a copy of the Package Insert, any periodic safety updates, and all other information as required by local regulation and/or the IRB/IEC. At the end of the study, the investigator must notify the IRB/IEC about the study's completion. The IRB/IEC also must be notified if the study is terminated prematurely. Finally, the investigator must report to the IRB/IEC on the progress of the study at intervals stipulated by the IRB/IEC.

Voluntary informed consent must be obtained in writing from every subject. The obtaining of consent shall be documented before any procedure specific to the clinical investigation is applied to the subject.

The investigator must have a defined process for obtaining the required consent. Specifically, the investigator, or their delegate, must explain the clinical study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The subject must be provided an opportunity to ask questions of the investigator, and if required by local regulation, other qualified personnel. The investigator must provide the subject with a copy of the consent form written in a language the subject understands. The consent document must meet all applicable local laws and provide subjects with information regarding the purpose, procedures, requirements, and restrictions of the study, along with any known risks and potential benefits associated with the IP and the study, the available compensation, and the established provisions for maintaining confidentiality of personal, protected health information. Subjects will be told about the voluntary nature of participation in the study and must be provided with contact information for the appropriate individuals should questions or concerns arise during the study. The subject also must be told that their records may be accessed by appropriate authorities and sponsor-designated personnel. The investigator must keep the original, signed copy of the consent (file in subject's medical records) and must provide a duplicate copy to each subject according to local regulations.

The study sponsor assures that the key design elements of this protocol will be registered on www.clinicaltrials.gov if required by current regulations and, if applicable, other public databases as required by local country regulations. In addition, results of this study will be made publicly available on www.clinicaltrials.gov regardless of outcome if required by current regulations and, if applicable, in other public databases as required by local country regulations.

#### 15 REFERENCES

## 15.1 Regulations and Standards

The following references may be applicable in whole or in part for this clinical trial.

- ISO 11980:2012 Ophthalmic optics Contact lenses and contact lens care products Guidance for clinical investigations
- EN ISO 14155:2020 Clinical investigation Investigation of medical devices Medical Devices for human subjects Human Subjects Good Clinical Practice

- 21 CFR Part 11 Electronic Records; Electronic Signatures
- 21 CFR Part 50 Protection of Human Subjects
- 21 CFR Part 56 Institutional Review Boards
- 21 CFR Part 812 Investigational Device Exemptions
- 21 CFR Part 54 Financial Disclosure by Clinical Investigators

## 15.2 Scientific and Other References

Not applicable. There are no references.







Signature Page for V-CLN-0010987 v5.0  $\,$